CLINICAL TRIAL: NCT01891669
Title: A PHASE 1, DOSE ESCALATION STUDY OF PF-06263507 IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study Of PF-06263507 In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on June 23, 2015 due to the company's change in prioritization for the portfolio and is not due to any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B4481001
Record Dates: First submitted 2013-06-10; First posted 2013-07-03 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Neoplasms; Carcinoma, Non Small Cell Lung; Breast Neoplasms; Ovarian Neoplasms
Keywords: ADC 5T4; PF-06263507; solid tumors; lung cancer; breast cancer; ovarian cancer; cancer; tumors; neoplasm metastasis
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Neoplasm Metastasis | interventions — PF-06263507

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Part 1 (Experimental)
  Interventions: Drug: PF-06263507

INTERVENTIONS:
Drug: PF-06263507 — Part 1 - PF-06263507 will be administered intravenously in 21-day cycles in cohorts of 2 or more patients starting at a dose of 0.05 mg/kg. Increases in dose will continue until MTD is determined.
Drug: PF-06263507 — Part 2 - Patients with select tumor types will be treated at the MTD or Recommended Phase 2 dose selected in Part 1.

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-06263507 in patients with advanced solid tumors in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of solid tumor that is advanced/metastatic and resistant to standard therapy or for which no standard therapy is available.
* Performance Status of 0 or 1.
* Adequate bone marrow, kidney, liver, and heart function.

Exclusion Criteria:

* Brain metastases requiring steroids.
* Major surgery or anti-cancer therapy within 4 weeks of study treatment start.
* Active bacterial, fungal or viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08-08 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2015-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Shapiro GI, Vaishampayan UN, LoRusso P, Barton J, Hua S, Reich SD, Shazer R, Taylor CT, Xuan D, Borghaei H. First-in-human trial of an anti-5T4 antibody-monomethylauristatin conjugate, PF-06263507, in patients with advanced solid tumors. Invest New Drugs. 2017 Jun;35(3):315-323. doi: 10.1007/s10637-016-0419-7. Epub 2017 Jan 9. PMID 28070718

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06263507 0.05 mg/kg: PF-06263507 0.05 mg/kg was administered on Day 1 of each 21-day cycle as an intravenous (IV) infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 0.1 mg/kg: PF-06263507 0.1 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 0.19 mg/kg: PF-06263507 0.19 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 0.37 mg/kg: PF-06263507 0.37 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 0.73 mg/kg: PF-06263507 0.73 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 1.42 mg/kg: PF-06263507 1.42 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 2.78 mg/kg: PF-06263507 2.78 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 4.34 mg/kg: PF-06263507 4.34 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 5.42 mg/kg: PF-06263507 5.42 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
- PF-06263507 6.5 mg/kg: PF-06263507 6.5 mg/kg was administered on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes. A cycle was defined as the time from Day 1 dose to the next Day 1 dose.
Period: Overall Study
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Completed | 0 | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 1
Not Completed | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (2.1) | 57 (4.2) | 41 (22.6) | 60 (7.1) | 53.5 (14.8) | 62 (36.8) | 61.5 (7.8) | 65.2 (9.9) | 57.7 (5.1) | 67.7 (5.9) | 59.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 4 | 2 | 1 | 15
  MALE | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: DLT was defined as any of the following adverse events (AEs) occurring in the first cycle of treatment (21 days) which were attributable to PF-06263507: 1) Grade 4 neutropenia lasting >7 days, 2) Febrile neutropenia, 3) Grade >=3 neutropenia with infection, 4) Any grade thrombocytopenia associated with clinically significant or life-threatening bleeding, 4) Grade 4 thrombocytopenia, 5) Any grade >=3 non-hematologic toxicities, 6) A positive cardiac troponin I result, 7) Persisting non-hematologic toxicities resulted in more than 2 weeks delay in receiving the next scheduled cycle. Severity of AEs was graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Baseline up to Cycle 2 Day 1 (22 days)
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), by Maximum National Cancer Institute (NCI) Common Terminology Criteria (CTC) for AEs (CTCAE) (Version 4.0) Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs are events which occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. If the same participant in a given treatment had more than 1 occurrence in the same preferred term event category, only the worst CTCAE grade was reported.
Time Frame: Baseline, Day 1 to 15 for Cycle 1, Day 1 to end of treatment for Cycle 2 and subsequent cycles, and follow-up.
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
participants
  Any AEs, Grade 1 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0
  Any AEs, Grade 2 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 1
  Any AEs, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2
  Any AEs, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any AEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any AEs, Total | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3

3. Secondary Outcome: Number of Participants With Treatment-related AEs, by Maximum NCI CTCAE (Version 4.0) Grade
Description: as for outcome 2
Time Frame: Baseline, Day 1 to 15 for Cycle 1, Day 1 to end of treatment for Cycle 2 and subsequent cycles, and follow-up.
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
participants
  Any AEs, Grade 1 | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 4 | 1 | 0
  Any AEs, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Any AEs, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Any AEs, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AEs, Total | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 6 | 3 | 3

4. Secondary Outcome: Number of Participants With Hematological Test Abnormalities in All Cycles.
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 hematological test abnormalities.
Time Frame: Baseline, Days 1, 3, 8 and 15 for Cycle 1, Days 1, 8, 15 for Cycle 2 and subsequent cycles, and end of treatment
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Participants
  Anemia Grade 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 4 | 1 | 2
  Anemia Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1
  Hemoglobin increased Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphopenia Grade 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 2
  Lymphopenia Grade 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0
  Lymphopenia Grade 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Lymphopenia Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets Grade 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0
  Platelets Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Platelets Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White blood cells (WBC) Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Chemistry Test Abnormalities in All Cycles.
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 chemistry tests abnormalities.
Time Frame: Baseline, Days 1, 3, 8 and 15 for Cycle 1, Days 1, 8, 15 for Cycle 2 and subsequent cycles, and end of treatment
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Participants
  Alanine aminotransferase (ALT) Grade 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 1
  Alkaline phosphatase Grade 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 3 | 1 | 1
  Alkaline phosphatase Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Alkaline phosphatase Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate aminotransferase (AST) Grade 1 | 1 | 1 | 2 | 0 | 1 | 1 | 2 | 4 | 0 | 1
  AST Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  AST Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Bilirubin (total) Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Bilirubin (total) Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine Grade 1 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 2 | 1
  Creatinine Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypercalcemia Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypercalcemia Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperglycemia Grade 1 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 5 | 1 | 1
  Hyperglycemia Grade 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Hyperkalemia Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Hypernatremia Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia Grade 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 1
  Hypoalbuminemia Grade 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2
  Hypocalcemia Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Hypocalcemia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypoglycemia Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypokalemia Grade 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 0
  Hypokalemia Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypomagnesemia Grade 1 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 3 | 1
  Hyponatremia Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 2
  Hyponatremia Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypophosphatemia Grade 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Hypophosphatemia Grade3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormalities in Urine Protein in All Cycles.
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 abnormalities in urine protein.
Time Frame: Baseline, Day 15 for Cycle 1, Day 1 for Cycle 2 and subsequent cycles, and end of treatment
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Participants
  Urine protein Grade 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine protein Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Categorical Summarization Criteria
Description: Criteria for potentially clinically important (PCI) change in vital signs included: sitting systolic blood pressure (SBP) of <90 millimeters of mercury (mm Hg) or change in sitting SBP of >=30 mm Hg, sitting diastolic blood pressure (DBP) of <50 mm Hg or change in sitting DBP of >=20 mm Hg, sitting pulse rate of <40 or >120 beats per minute (bpm).
Time Frame: Baseline, Days 1, 3, 8 and 15 for Cycle 1, Days 1, 8, 15 for Cycle 2 and subsequent cycles, end of treatment, and follow-up.
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Participants
  DBP <50 mm Hg | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SBP maximum increase from baseline >=30 mm Hg | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
  DBP maximum increase from baseline >=20 mm Hg | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
  SBP maximum decrease from baseline >=30 mm Hg | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1
  DBP maximum decrease from baseline >=20 mm Hg | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0

8. Secondary Outcome: Number of Participants With Positive Anti-PF-06263507 Antibody
Description: The number of participants with positive anti-PF-06263507 antibody.
Time Frame: Pre-dose Day 1, Cycle 1 Day 15, Day 1 of every Cycle, up to 21 days after the last dose of study medication
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Participants | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: Number of participants with best overall response. Complete response (CR)=disappearance of all target lesions. Partial Response (PR)>=30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions. Progressive disease (PD) >=20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of the longest dimensions since treatment start, or the appearance of >=1 new lesion. Stable disease (SD)=neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months.
Population: Participants who had received at least one dose of study medication and had a baseline tumor assessment
Measure: Number; unit: pariticpants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
pariticpants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable/No response | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Objective progression | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 4 | 3 | 1
  Symptomatic deterioration | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Early death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Interminate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1

10. Secondary Outcome: Objective Response
Description: Number of particpants with objective response: confirmed CR or confirmed PR according to RECIST. CR was defined as the disappearance of all target lesions. A PR was defined as a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. To be assigned a status of PR or CR, changes in tumor measurements in participants with responding tumors had to have been confirmed by repeat studies that were performed ≥ 4 weeks after the criteria for response were first met.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months.
Population: Participants who had received at least one dose of study medication and had a baseline tumor assessment
Measure: Number; unit: pariticpants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
pariticpants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from initial dose until death from any cause, and was measured in the intent-to-treat population.
Time Frame: Baseline to death
Population: All enrolled participants
Measure: Number; unit: pariticpants
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
pariticpants
  Number of deaths | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Number for censored | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 5 | 3 | 2

12. Secondary Outcome: Time to Reach Maximum Observed Serum PF-06263507 Concentration (Tmax)
Time Frame: Baseline,Cycle 1 Day 1 pre-dose,1,4,8,12,24, and 48 hrs post dose,Day 5,Day 8 and Day 15;Day 1 of Cycle 2 and 3,Day 1 of Cycle 4 pre-dose,1,8,12,24 hr post dose, Day 8 and Day 15,every cycle thereafter on day 1 pre-dose, and up to 21 days after last dose.
Population: All enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
hour | 1.07 [1.03 to 1.10] | 1.00 [1.00 to 1.00] | 2.49 [0.983 to 4.00] | 1.01 [1.00 to 1.02] | 1.03 [1.02 to 1.03] | 1.02 [1.00 to 1.03] | 2.49 [1.00 to 3.98] | 1.13 [0.983 to 11.0] | 1.03 [1.00 to 1.03] | 1.22 [1.17 to 7.93]

13. Secondary Outcome: Time to Reach Maximum Observed Serum PF-06281192 Concentration (Tmax)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
hour | 1.07 [1.03 to 1.10] | 4.00 [4.00 to 4.00] | 2.53 [1.05 to 4.00] | 1.01 [1.00 to 1.02] | 6.01 [1.02 to 11.0] | 1.02 [1.00 to 1.03] | 7.44 [3.98 to 10.9] | 4.00 [1.07 to 8.08] | 8.00 [1.03 to 8.05] | 3.90 [1.17 to 4.02]

14. Secondary Outcome: Time to Reach Maximum Observed Serum PF-06264490 Concentration (Tmax)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 3 | 3
hour | 36.2 [24.4 to 48.0] | 16.0 [8.00 to 24.0] | 37.2 [26.3 to 48.0] | 51.0 [4.00 to 98.0] | 9.99 [7.98 to 12.0] | 9.51 [8.12 to 10.9] | 8.02 [7.30 to 12.0] | 8.13 [8.05 to 70.8] | 8.25 [7.93 to 8.28]

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment/withdrawal
Arm/Group | PF-06263507 0.05 mg/kg | PF-06263507 0.1 mg/kg | PF-06263507 0.19 mg/kg | PF-06263507 0.37 mg/kg | PF-06263507 0.73 mg/kg | PF-06263507 1.42 mg/kg | PF-06263507 2.78 mg/kg | PF-06263507 4.34 mg/kg | PF-06263507 5.42 mg/kg | PF-06263507 6.5 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 1/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 2/2 | 2/2 | 2/2 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06263507 0.05 mg/kg (N=2) | PF-06263507 0.1 mg/kg (N=2) | PF-06263507 0.19 mg/kg (N=2) | PF-06263507 0.37 mg/kg (N=2) | PF-06263507 0.73 mg/kg (N=2) | PF-06263507 1.42 mg/kg (N=2) | PF-06263507 2.78 mg/kg (N=2) | PF-06263507 4.34 mg/kg (N=6) | PF-06263507 5.42 mg/kg (N=3) | PF-06263507 6.5 mg/kg (N=3)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06263507 0.05 mg/kg (N=2) | PF-06263507 0.1 mg/kg (N=2) | PF-06263507 0.19 mg/kg (N=2) | PF-06263507 0.37 mg/kg (N=2) | PF-06263507 0.73 mg/kg (N=2) | PF-06263507 1.42 mg/kg (N=2) | PF-06263507 2.78 mg/kg (N=2) | PF-06263507 4.34 mg/kg (N=6) | PF-06263507 5.42 mg/kg (N=3) | PF-06263507 6.5 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal deposits (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation decreased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 4 | 2 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Waist circumference increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated prematurely before treatment in Part 2 started due to a business-related decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.